CLINICAL TRIAL: NCT00429923
Title: A Phase 3 Multicenter, Randomized, Double-Masked, Placebo-Controlled Study of the Safety and Efficacy of Difluprednate in the Treatment of Inflammation Following Ocular Surgery
Brief Title: Study of Difluprednate in the Treatment of Inflammation Following Ocular Surgery (ST-601A-002a)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sirion Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ST-601A-002a
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Results first posted 2009-07-02 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-05

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — difluprednate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Difluprednate 0.05% BID (Experimental): Difluprednate 0.05% 1 drop BID for 14 days.
  Interventions: Drug: Difluprednate
- Difluprednate 0.05% QID (Experimental): Difluprednate 0.05% 1 drop QID for 14 days.
  Interventions: Drug: Difluprednate
- Placebo (Placebo Comparator): Placebo for 14 days. Placebo was administered BID for 14 days and QID for 14 days. The outcomes of the 2 placebo groups were examined and were determined to be statistically indistinguishable so the placebo groups were pooled for comparison with the difluprednate groups.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Difluprednate
  Arms: Difluprednate 0.05% BID
Drug: Difluprednate
  Arms: Difluprednate 0.05% QID
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this phase III study is to determine the efficacy of difluprednate in the treatment of inflammation following ocular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral ocular surgery in the day prior to study enrollment.
* Anterior chamber cell grade ≥ "2" on the day after surgery (Day 1).
* Aged 2 years or older on the day of consent.
* Negative urine pregnancy test on Day 1 for postmenarchal subjects; negative urine pregnancy test for premenarchal subjects at the investigator's discretion.
* Provide signed written consent prior to entering the study or signed written consent from parent or legal guardian if subject is a minor and signed assent from minor subject, if appropriate.

Presurgical Exclusion Criteria:

* Systemic administration of any corticosteroid in the 2 weeks prior to study enrollment.
* Periocular injection in the study eye of any corticosteroid solution within 4 weeks prior to instillation of the study drug, or of any corticosteroid depot within 2 months prior to instillation of the study drug.
* Instillation of any topical ocular corticosteroid or NSAID within 24 hours prior to instillation of the study drug or during the course of the study, with the exception of presurgical administration of a topical NSAID to prevent miosis.
* Any history of glaucoma or ocular hypertension in the study eye.
* History or presence of endogenous uveitis.
* Any current corneal abrasion or ulceration.
* Any confirmed or suspected active viral, bacterial, or fungal keratoconjunctival disease.
* Allergy to similar drugs, such as other corticosteroids.
* History of steroid-related IOP increase.
* Scheduled surgery on the contralateral eye during the treatment period.
* Unwilling to discontinue use of contact lenses during the study period.
* Pregnancy or lactation.
* Participation in any study of an investigational topical or systemic new drug or device within 30 days prior to screening, or at any time during the study.
* Prior participation in the study described in this protocol.
* Unable or unwilling to give signed informed consent prior to participation in any study related procedures.

Postsurgical Exclusion Criteria:

* Ocular hemorrhage which interferes with evaluation of postsurgery inflammation.
* Injection of gas into the vitreous body during surgery.
* Presence of IOP ≥24 mm Hg on Day 1 after surgery.

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 219 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Vogel, MD, Study Chair — Sirion Therapeutics, Inc.
Locations (1):
- Comprehensive Eye Care, Washington, Missouri, United States

REFERENCES:
- [Derived] Korenfeld MS, Silverstein SM, Cooke DL, Vogel R, Crockett RS; Difluprednate Ophthalmic Emulsion 0.05% (Durezol) Study Group. Difluprednate ophthalmic emulsion 0.05% for postoperative inflammation and pain. J Cataract Refract Surg. 2009 Jan;35(1):26-34. doi: 10.1016/j.jcrs.2008.09.024. PMID 19101421

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled February 6, 2007 and last subject completed September 17, 2007 at 13 sites in the United States.
Pre-assignment Details: Subjects enrolled if, 24 hours after ocular surgery, they had an anterior chamber cell grade of ≥ "2" and met the protocol inclusion and exclusion criteria.
Period: Overall Study
Arm/Group | Difluprednate 0.05% BID | Difluprednate 0.05% QID | Placebo
Started | 57 | 55 | 107
Completed | 52 | 51 | 68
Not Completed | 5 | 4 | 39
Not completed — Adverse Event | 0 | 2 | 3
Not completed — Lack of Efficacy | 4 | 1 | 33
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Withdrew Consent | 1 | 0 | 1
Not completed — Early Termination | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Difluprednate 0.05% BID | Difluprednate 0.05% QID | Placebo | Total
Number analyzed (Participants) | 57 | 55 | 107 | 219
Age Continuous [Mean (Standard Deviation); unit: years] | 70.8 (0) | 68.1 (0) | 69.1 (0) | 69.3 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 51 | 112.0
  Male | 27 | 24 | 56 | 107.0

OUTCOME MEASURES:

1. Primary Outcome: Anterior Chamber Cell Grade of "0" on Day 8 (Difluprednate QID vs Placebo).
Description: Measured on a 0 to 4 scale: "0" is ≤ 1 cell; "1" is 2-10 cells; "2" is 11-20 cells; "3" is 21-50 cells; "4" is > 50 cells.
Time Frame: Day 8 (QID)
Population: The ITT population was defined as all randomized subjects who received at least 1 administration of the study drug. Analysis of the ITT population, with LOCF for missing data, was conducted for all primary and secondary endpoints at Days 3, 8, 15, and 29.
Measure: Number; unit: participants
Arm/Group | Difluprednate 0.05% BID | Difluprednate 0.05% QID | Placebo
Number analyzed (Participants) | 0 | 55 | 105
participants
  Proportion of subjects w/AC cell grade=0 on Day 8 | 0 | 19 | 13
Statistical Analysis 1: Comparison: Difluprednate 0.05% QID vs Placebo; Test type: Superiority or Other; p = 0.0014, Mantel Haenszel

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days